CLINICAL TRIAL: NCT06270277
Title: Evaluation of Quality of Life and Psychosocial Status in Children With Inflammatory Bowel Disease: Prospective Controlled Trial
Brief Title: Evaluation of Quality of Life and Psychosocial Status in Children With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Busra Tetik Dincer, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 30.01.2024-4272
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Diseases; Psychosocial Impairment
Keywords: Inflammatory bowel diseases; Psychosocial condition; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Adolescents with Inflammatory bowel diseases and healthy control group in same age will be administered Pediatric Quality of Life Inventory (PedsQL) and Strengths and Difficulties Questionnaire (SDQ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflammatory bowel disease group (Experimental): Adolescents with Inflammatory bowel diseases will be administered Pediatric Quality of Life Inventory (PedsQL) and Strengths and Difficulties Questionnaire (SDQ).
  Interventions: Diagnostic Test: Pediatric Quality of Life Inventory (PedsQL); Diagnostic Test: Strengths and Difficulties Questionnaire (SDQ)
- Control group (Active Comparator): Adolescents without known diseases in same age group will be administered Pediatric Quality of Life Inventory (PedsQL) and Strengths and Difficulties Questionnaire (SDQ) as control group
  Interventions: Diagnostic Test: Pediatric Quality of Life Inventory (PedsQL); Diagnostic Test: Strengths and Difficulties Questionnaire (SDQ)

INTERVENTIONS:
Diagnostic Test: Pediatric Quality of Life Inventory (PedsQL) — Questionnaire
Diagnostic Test: Strengths and Difficulties Questionnaire (SDQ) — Questionnaire

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic condition that affects the psychosocial status and physical activities of children and their parents in many ways. Our study aimed to investigate the variability of disease-related quality of life and behavioral and emotional adjustment issues compared to a healthy control group among adolescents and their families diagnosed with IBD. Children with IBD and the healthy control group, as well as the parents of both groups, will administered the Pediatric Quality of Life Inventory (PedsQL) and Strengths and Difficulties Questionnaire (SDQ). The PedsQL is a scale used to assess physical and psychosocial functioning based on the individual's own experiences, commonly employed in clinical trials and quality improvement initiatives. The scale evaluates physical activity status and psychosocial functioning through questions related to emotional, social, and school-related issues.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8-17 years
* Diagnosed Inflammatory bowel disease
* Healthy adolescents aged between 8-17 years

Exclusion Criteria:

* Not obtaining informed consent
* Diagnosis of psychiatric disorder

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) score | 1 day after questionnaire
  Score of questionnaire
Strengths and Difficulties Questionnaire (SDQ) | 1 day after questionnaire
  Score of questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nafiye Urgancı, M.D., Study Director — Sisli Hamidiye Etfal Training and Research Hospital, Division of pediatric gastroenterology
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No